CLINICAL TRIAL: NCT01109914
Title: Immune Response After Inactivated Oral Cholera Vaccine (Dukoral) in Renal Transplant Recipients
Brief Title: Mucosal Response in Immunocompromised Host
Acronym: MICH
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Leiden University Medical Center (Other)
Collaborators: Crucell B.V., Leiden, the Netherlands (Unknown)
Responsible Party: Principal Investigator, Darius Soonawala, Drs, Leiden University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MICH P10.011
Record Dates: First submitted 2010-04-22; First posted 2010-04-23 (Estimated); Last update posted 2015-03-26 (Estimated); Status verified 2015-03

CONDITIONS: Kidney Transplantation; Immunity
Keywords: Renal transplantation; Immunosuppression; ETEC; Dukoral; Vaccination; Immunity, Humoral
MeSH Terms: interventions — Dukoral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Renal transplant recipients (MMF) (Experimental): Renal transplant recipients using prednisolone and mycophenolate mofetil (MMF) but no other immunosuppressive drug.
  Intervention: vaccination with Dukoral
  Interventions: Biological: Dukoral
- Renal transplant recipients (CNI) (Experimental): Renal transplant recipients using prednisolone and a calcineurin inhibitor (cyclosporine or tacrolimus) but no other immunosuppressive drug.
  Intervention: vaccination with Dukoral
  Interventions: Biological: Dukoral
- Healthy volunteers (Experimental): Healthy volunteers (partners, brothers or sisters of the renal transplant recipients).
  Intervention: vaccination with Dukoral
  Interventions: Biological: Dukoral

INTERVENTIONS:
Biological: Dukoral — Two oral doses of Dukoral® (SBL Vaccines) will be administered (day 0 and day 14). Each dosage contains 3 ml of suspension in a vial and 5.6 g of effervescent granules in a sachet. Each dosage (3 ml) contains: A total of 100000 million bacteria of the following strains:
  * Vibrio cholerae O1 Inaba, classical biotype (heat inactivated) 25x1000 million bacteria*
  * Vibrio cholerae O1 Inaba, El Tor biotype (formalin inactivated) 25x1000 million bacteria*
  * Vibrio cholerae O1 Ogawa, classical biotype (heat inactivated) 25x1000 million bacteria*
  * Vibrio cholerae O1 Ogawa, classical biotype (formalin inactivated) 25x1000 million bacteria*
  * Recombinant cholera toxin B subunit (rCTB) 1 mg (produced in V. cholerae O1 Inaba, classical biotype strain 213)

SUMMARY:
The aim of this study is to verify whether vaccination with Dukoral® (SBL Vaccines) induces an immune response in renal transplant recipients on prednisolone in combination with either a calcineurin inhibitor CNI) or mycophenolate mofetil (MMF).

DETAILED DESCRIPTION:
BACKGROUND:

LT-ETEC is the most common cause of travelers' diarrhoea. Dukoral® (SBL Vaccines) reduces the severity and duration of LT-ETEC induced diarrhea. Dehydration due to diarrhea poses a risk to the health of renal transplant recipients. Therefore Dukoral may benefit this group of travelers.

AIM OF THIS STUDY:

Primary objective: To verify whether vaccination with Dukoral® (SBL Vaccines) induces an immune response in renal transplant recipients on prednisolone in combination with either a calcineurin inhibitor (cyclosporine or tacrolimus) or mycophenolate mofetil.

Secondary objective: To evaluate to what extent, the immune response differs, depending on the use of different classes of immunosuppressive drugs (CNI or MMF).

STUDY DESIGN:

Single center interventional study.

Population: The population base of the study consists of adult renal transplant recipients who received their transplant at our medical center. The control population consists of the healthy partners and siblings of the renal transplant recipients. We intend to include 10 healthy volunteers and 60 renal transplant recipients (20 on prednisolone and a CNI and 20 on prednisolone and MMF).

Intervention: Dukoral® (SBL Vaccines) will be administered orally at baseline (day 0) and at day 14.

Laboratory analysis: Serum CTB antibody (ELISA), Vibriocidal assay. The analysis is performed at Crucell.

Statistical analysis: No formal sample-size calculation was performed. The crude outcome estimates will be adjusted for variables that may influence the outcome (age, time after transplantation, past treatment for transplant rejection, current renal function, cumulative prednisolone dose, serum concentration (i.e. area under the curve) of CNI and MMF.

Note: the study intended to also recruit a study arm consisting of patients on a mTORi. Recruitment for this study arm was unsuccesful due to the scarcity of elligible patients.

ELIGIBILITY:
HEALTHY VOLUNTEERS

Inclusion criteria:

* Above 18 years of age
* Informed consent

Exclusion Criteria:

* History of an auto-immune disease (SLE, ANCA associated vasculitis, Goodpasture, Henoch Schonlein, cryoglobulinemia, secondary vasculitis, polyarteritis nodosa and immunodeficiency disorders like IgA deficiency)
* Chronic infection
* Past vaccination with Dukoral or another cholera or ETEC vaccine
* History of infection with Vibrio cholerae
* Episode of diarrhoea in the 6 months prior to inclusion
* Allergy to vaccine-specific components
* History of a severe allergic reaction to any vaccine
* Treatment with blood products in the 3 months prior to inclusion
* Current pregnancy or breastfeeding
* Premenopausal women not willing to use contraceptives during the first 60 days after vaccination
* Use of any immunosuppressive drug

RENAL TRANSPLANT RECIPIENTS

Inclusion Criteria:

* Above 18 years of age
* Creatinin clearance ≥ 40 ml/min measured in the 6 months prior to inclusion
* Stable renal function for 1 year prior to inclusion
* Stable immunosuppressive regimen of a CNI, MMF or mTORi combined with prednisolone for at least 3 months prior to inclusion
* Informed Consent

Exclusion Criteria:

* History of an auto-immune disease (SLE, ANCA associated vasculitis, Goodpasture, Henoch Schonlein, cryoglobulinemia, secondary vasculitis, polyarteritis nodosa and immunodeficiency disorders like IgA deficiency)
* Chronic infection
* Treatment for rejection of the transplant in the past 1 year prior to inclusion
* Past vaccination with Dukoral or another cholera or ETEC vaccine
* History of infection with Vibrio cholerae
* Episode of diarrhoea in the 6 months prior to inclusion
* Allergy to vaccine-specific components
* History of a severe allergic reaction to any vaccine
* Treatment with blood products in the 3 months prior to inclusion
* Current pregnancy or breastfeeding
* Premenopausal women not willing to use contraceptives during the first 60 days after vaccination
* Use of an immunosuppressive drug other than CNI, MMF, mTORi or prednisolone at the the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage seroconversion among all renal transplant recipients. | day 20-22
  ≥3-fold rise in serum anti-CTB antibodies or ≥4-fold rise in serum vibriocidal antibodies.

SECONDARY OUTCOMES:
Group differences in geometric mean antibody titers after vaccination | day 20-22
  post-vaccination anti-rCTB titers, measured by Enzyme Immuno Assay (EIA); post-vaccination serum vibriocidal antibodies, measured in vibriocidal assay.

CONTACTS AND LOCATIONS:
Overall Officials: Leo G Visser, MD PhD, Principal Investigator — Leiden University Medical Center; Darius Soonawala, MD, Study Director — Leiden University Medical Center; O W Bredewold, MD, Study Chair — Leiden University Medical Center; J W de Fijter, Prof PhD, Study Chair — Leiden University Medical Center; Marjolein AC Uijlings, Study Chair — Leiden University Medical Center; Emile FF Jonker, MD, Study Chair — Leiden University Medical Center
Locations (1):
- Leiden Univeristy Medical Centre, Leiden, South Holland, Netherlands

REFERENCES:
- [Derived] Jonker EFF, Uijlings MAC, Visser LG, Soonawala D. Comparison of the immunogenicity of Dukoral(R) oral cholera vaccine between renal transplant recipients on either a calcineurin inhibitor or mycophenolate - A controlled trial. Vaccine. 2019 May 21;37(23):3133-3139. doi: 10.1016/j.vaccine.2019.04.010. Epub 2019 Apr 24. PMID 31029516